CLINICAL TRIAL: NCT00838851
Title: Range of Neutrophil Response to 20,000 EU of Clinical Center Reference Endotoxin in Normal Adult
Brief Title: Response of Airway Cells to 20,000 EU of Endotoxin in Normal Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: no further funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, David B. Peden, MD, Professor of Pediatrics, Director of CEMALB, University of North Carolina, Chapel Hill
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 03-1523 (GCRC 2040); 1RC1ES018417 (NIH)
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Controls
Keywords: endotoxin; CCRE; LPS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CCRE (Experimental)
  Interventions: Biological: Clinical Center Reference Endotoxin (CCRE)

INTERVENTIONS:
Biological: Clinical Center Reference Endotoxin (CCRE) — Inhalation of 20,000 EU Clinical Center Reference Endotoxin (CCRE)
  Other Names: LPS

SUMMARY:
The purpose of this study is to determine the range of neutrophil response (influx of PMNs to the airways as determined in sputum) after inhalation of CCRE (20,000 EU).

DETAILED DESCRIPTION:
Twenty-four or forty-eight hours (study day 1) prior to the inhalation challenge, subjects will undergo a physical examination of the ears, nose, throat and chest and will have an assessment of vital signs (temperature, pulse, respiratory rate, blood pressure), oxygen saturation, symptom score assessment and undergo spirometry to rule out acute illness prior to challenge. All female volunteers will undergo a urine pregnancy test. A similar examination will take place immediately prior to inhalation challenge with 20,000 EU of CCRE, as well as 30, 60, 120, 180, 240, 300 and 360 minutes and 24 hours after challenge (with the exception of a pregnancy test which will only be administered prior to sputum induction on study day 1). Induced sputum will be 24 to 48 hours prior to challenge, and again six hours after challenge on Study day 2. Sputum will be analyzed for PMN content, CD14 expression on airway macrophages and monocytes, soluble CD14 levels, cytokine levels in sputum and products of inflammatory cells (eosinophil, cationic protein, myeloperoxidase). Blood will be collected for a CBC and differential when the pre- challenge induced sputum is obtained and again 6 hours after challenge and 24 hours after challenge. Blood lymphocytes from a 10 ml aliquot will be assessed for lymphocyte subset and activation markers, as well as proliferative and cytokine responses. Blood will also be collected and will be assessed by whole blood assays for markers of inflammatory and immune activation (CD11b, CD14, CD64, CD16, HLA-DR, CD45, CD3, CD80, CD86, CD83, CD40) and function (phagocytosis and oxidative burst) by three color flow cytometry. Plasma will be separated from 4 ml and frozen at 70° C for future analysis of mediators of interest, such as cytokines, as well as other systemic effects of endotoxin.

Subjects will then be discharged to home with contact information for study staff. If a volunteer has an unexpected complication such as shortness of breath, decrease in pulmonary function, unstable vital signs or other he or she will be admitted to the GCRC for overnight observation. The next morning (study day 3) subjects will return to the CEMALB for a final set of vital signs, spirometry, symptom scoring, a venipuncture and an examination by a study physician.

Each volunteer will be given a symptom scoring sheet for each day up to 96 hours (4 days) after challenge.

Each sheet will include the name and phone number of the study coordinator and study MD. Sample home symptom scoring sheets and instructions are included with this protocol.

Between 48 and 96 hours after challenge, each volunteer will be called to determine their status, inquiring about symptoms, symptom scoring, and need for medication and/or physician visits.

Between 7 and 10 days of the challenge dose, each subject will be asked to return for a study discontinuation visit. At that time temperature, pulse, systolic and diastolic BP, respiratory rate, FVC and FEV1 and SpO2 (oxygen saturation), and symptoms scores will be assessed and, if abnormal, medical evaluation as directed by the study physician will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion: Healthy, non-allergic, non-asthmatic 18-50 year old males and females with a < 0.5 pack year history of tobacco use who have a negative allergy skin test, normal lung function, defined as (Knudsen 1976/1984 predicted set):

  1. FVC of > 80 % of that predicted for gender, ethnicity, age and height
  2. FEV1 of > 80 % of that predicted for gender, ethnicity, age and height
  3. FEV1/FVC ratio of > 75% of that predicted for gender, ethnicity , age and height
* Oxygen saturation of > 94 %,
* Normal blood pressure (Systolic between 150 - 90, Diastolic between 90-60 mm Hg),
* Symptom Score no greater than 6 (out of a possible 24) for total symptom score with a value no greater than 2 for any one score. No score may be greater than 2,
* Negative methacholine inhalation challenge.
* On the day of a challenge, body temperature must be no greater than 37.8 degrees, measured orally.

Exclusion Criteria:

* A history of significant chronic illnesses (to include diabetes, autoimmune diseases, immunodeficiency state, known ischemic heart disease, chronic respiratory diseases such as chronic obstructive pulmonary disease or asthma, hypertension).
* Allergy to any medications which may be used in the course of this study (albuterol, acetaminophen, aspirin or non-steroidal anti-inflammatory agents, corticosteroids, lactose).
* Positive pregnancy test within 48 hours of the time of challenge.
* Medications which may impact the results of the endotoxin challenge, interfere with any other medications potentially used in the study (to include steroids, beta antagonists, non-steroidal anti-inflammatory agents) or suggest an ongoing illness (such as antibiotics).
* Acute, non-chronic, medical conditions, including (but not limited to) pneumonia or bronchitis requiring antibiotics, febrile illnesses, flu-like symptoms must be totally resolved symptomatically for 2 weeks.
* Unspecified illnesses, which in the judgment of the investigator increase the risk associated with endotoxin inhalation challenge, will be a basis for exclusion.
* Persons employed within the past 6 months in an occupation with high risk for endotoxin exposure (specifically persons working in a swine confinement facility, cotton storage or grain storage site)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2003-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Neutrophil response (influx of PMNs to the airways as determined in sputum) after inhalation of CCRE (20,000 EU), | 0-24 hours post challenge

SECONDARY OUTCOMES:
changes in PFT's and vital signs | 0-21 days post challenge

CONTACTS AND LOCATIONS:
Overall Officials: David B Peden, MD, MS, Principal Investigator — University of North Carolina at Chapel Hill, Dept of Pediatrics / Center for Environmental Medicine, Asthma and Lung Biology
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States